CLINICAL TRIAL: NCT04587362
Title: The Diagnostic Ultrasound Enthesitis Tool (DUET) Study: Development of a Sonographic Enthesitis Score for Early Diagnosis of Psoriatic Arthritis
Brief Title: The Diagnostic Ultrasound Enthesitis Tool (DUET) Study
Acronym: DUET
Status: Completed | Type: Observational
Sponsor: Women's College Hospital (Other)
Collaborators: Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (Network)
Responsible Party: Sponsor
Other Study IDs: 2019-0194-B
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Psoriatic Arthritis; Psoriasis; Non-Inflammatory Rheumatic Conditions
Keywords: Enthesitis; PsA; Musculoskeletal Ultrasound; Diagnosis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psoriatic Arthritis: Subjects newly diagnosed with psoriatic arthritis (< 5 years), confirmed by a rheumatologist and fulfilling the ClASsification for Psoriatic ARthritis (CASPAR) criteria.
  Interventions: Diagnostic Test: Musculoskeletal Ultrasound
- Psoriasis without musculoskeletal symptoms: Patients with dermatologist confirmed psoriasis, without any history of Psoriatic Arthritis, and musculoskeletal symptoms.
  Interventions: Diagnostic Test: Musculoskeletal Ultrasound
- Non-Inflammatory Rheumatic conditions: Patients with non-inflammatory rheumatic conditions such as osteoarthritis, non-specific back pain, soft tissue rheumatism, degenerative tendinopathy and fibromyalgia. Patients with present or past history of psoriasis, psoriatic arthritis, known or suspected rheumatic inflammatory conditions (e.g. rheumatoid arthritis, spondyloarthritis and gout), and/or inflammatory bowel disease will be excluded.
  Interventions: Diagnostic Test: Musculoskeletal Ultrasound

INTERVENTIONS:
Diagnostic Test: Musculoskeletal Ultrasound — High quality ultrasound scanners and high-resolution transducers, will be used to scan 16 joints sites for each subject. Ultrasound had excellent spatial resolution, making it an highly efficient, non-invasive tool for the assessment on enthesitis, which is an early feature of psoriatic arthritis. It is an affordable and accessible tool that is widely used in rheumatology practice.

SUMMARY:
Psoriatic arthritis (PsA) is a type of joint disease that can lead to severe joint damage and disability within the first few years of the disease. This is why early detection and treatment of the disease is essential to prevent serious joint damage and improve long-term outcomes in these patients. However, there is currently no reliable way to tell the difference between PsA and other types of joint disease. This makes it difficult to detect PsA early. Enthesitis is an inflammation of the area where muscle tendons and ligaments attach to bones. Enthesitis is a key feature in PsA and can be easily detected using ultrasonography. The aim of this research study is to develop a system to evaluate enthesitis using ultrasonography, which can be used as an effective tool in the early detection of PsA. This will help in providing patients with early treatment to prevent further joint damage.

ELIGIBILITY:
General Inclusion Criteria:

* Age ≥18
* Able to provide an informed consent

Specific Inclusion Criteria for PsA:

* Meets the CASPAR criteria for PsA
* Early PsA - Less than 5 years from a rheumatologist diagnosis of PsA

Specific Inclusion Criteria for Psoriasis:

* Dermatologist confirmed diagnosis of psoriasis
* No prior diagnosis of PsA or signs of PsA on physical examination
* Psoriasis Epidemiology Screening Tool (PEST) score < 3

Specific Inclusion Criteria for non-inflammatory rheumatic disease:

* Referred to rheumatology for musculoskeletal symptoms such as joint pain, stiffness, back pain
* No evidence of inflammatory rheumatic condition including rheumatoid arthritis, spondyloarthritis, systemic lupus erythematosus, scleroderma, gout, septic arthritis or recent joint trauma/surgery
* No psoriasis
* No inflammatory bowel disease

Exclusion Criteria:

* Using any biologic medications including Tumor Necrosis Factor (TNF) inhibitors, Interleukin (IL)-17 inhibitors, IL-23 inhibitors, IL-12/23 inhibitors, Janus Kinase (JAK) inhibitors
* Prednisone ≥ 7.5 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited form rheumatology and dermatology clinics at participating recruitment sites throughout the world.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
DUET scoring system for early diagnosis of PsA | From beginning to end of physical & ultrasound assessment, up to 1.5 hours
  To derive the DUET scoring system for distinguishing PsA from non-inflammatory disease using musculoskeletal ultrasound. The investigators will report the optimal set of weighted parameters and their performance measures (area under the curve, suggested cut-off points, sensitivity, and specificity).

SECONDARY OUTCOMES:
Assess the construct validity of the new DUET scoring system | From beginning to end of physical & ultrasound assessment, up to 1.5 hours
  Construct validity of the newly derived DUET scoring system will evaluate its correlation with clinical measures of disease activity (e.g. total enthesitis count, joint count) and patient reported outcomes.
  The investigators will evaluate the agreement between central and local readers using the new scoring system to evaluate its reliability among local readers using intra-class correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Lihi Eder, MD, PhD, Principal Investigator — University of Toronto; Sibel Z Aydin, MD, Principal Investigator — University of Ottawa; Gurjit S Kaeley, MD, Principal Investigator — University of Florida
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Development and Validation of a Sonographic Enthesitis Instrument in Psoriatic Arthritis: The Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA) Diagnostic Ultrasound Enthesitis Tool (DUET) Project — http://pubmed.ncbi.nlm.nih.gov/32482769/